CLINICAL TRIAL: NCT05351268
Title: Safety and Efficacy of 3D Printing Coplanar Template Combined With CT Guided Radioactive I-125 Seed Implantation in the Treatment of Thoracic Malignant Tumors
Brief Title: 3DPCT Combined With CT Guided RISI in the Treatment of Thoracic Malignant Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BYSY-2022-3DPCT-TC
Record Dates: First submitted 2022-04-20; First posted 2022-04-28 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Radioactive Iodine-125 Brachytherapy; Thoracic Cancer; 3D Printing Coplanar Template; Nuclear Radiation Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3DPCT and CT guided RISI (Experimental): All patients were treated with clinical routine treatment: 3DPCT combined with CT guided radioactive seed implantation. Collect patient information and treatment information for analysis.
  Interventions: Radiation: Radioactive seed brachytherapy

INTERVENTIONS:
Radiation: Radioactive seed brachytherapy — The radioactive Iodine-125 seed can release low dose of irradiation persistently which kills tumors cell and causes less damage to normal tissue at the same time. The treatment was performed under CT monitoring. 3D-printing coplanar template includes information on the path of the implantation needle, the needle path can be controlled accurately which can make the operation more accurate.

SUMMARY:
The main technical difficulties in radioactive iodine-125 seed implantation (RISI) lie in the complexity of operation and the control of operation quality. The current data shows that under the combined guidance of 3D-printing template and CT, the accuracy of RISI has been significantly improved, and the actual target dose could meet the design requirements of preoperative plan.

At present, 3D printing templates (3DPT) are divided into non-coplanar templates (3DPNCT) and coplanar templates (3DPCT). In clinical practice, due to the complex technical requirements, high production cost and long printing time of 3DPNCT, a considerable number of patients can also complete the treatment with 3DPCT. Moreover, compared with 3DPNCT, 3DPCT has the advantages of accurate needle path control, fast needle path adjustment, convenient for intraoperative real-time optimization, without waiting for printing time, easy for doctors to master, lower cost than 3DPNCT, and easy to carry out at the grass-roots level. Therefore, this study intends to explore 3DPCT technology to further clarify: (1) the accuracy of 3DPCT assisted CT guided RISI in the treatment of thoracic malignant tumors; (2) the short-term efficacy and toxicity of 3DPCT assisted CT guided RISI in the treatment of thoracic malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of malignant tumor of chest, lesion diameter less than 7 cm.
* There is no extensive systemic metastasis or although there is metastasis, the metastasis have been controlled by early treatment.
* No bleeding tendency, anticoagulant therapy and / or antiplatelet coagulation drugs should be stopped for at least 1 week before treatment.
* No serious or uncontrolled underlying diseases (such as severe or uncontrolled hypertension, diabetes, cardiovascular and cerebrovascular diseases and organ dysfunction) are found.
* There is a suitable puncture path, and the therapeutic dose is expected to be achieved.
* KPS > 70, expected to tolerate puncture / seed implantation, and expected survival time greater than 3 months.

Exclusion Criteria:

* Severe impairment of lung function (such as FEV1 < 40% predicted value, FVC < 50% predicted value, DLCO < 40% predicted value).
* High risk of skin invasion and ulceration at the puncture site before treatment.
* There is a large range of liquefaction and necrosis in the lesion, and the expected seed distribution would be poor.
* Pregnant women, lactating women and mentally ill patients.
* The patient with poor compliance and unable to complete the treatment.
* Other conditions of the researchers who think it is not suitable to participate in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Local progression free survival | From the beginning of the treatment to 2 years after the treatment.
  The time from the date of SBRT to the date of local recurrence or death or the date of last observation.
Incidence of adverse events | From the beginning of the treatment to 2 years after the treatment.
  The adverse events are evaluated by the common terminology criteria for adverse events (CTCAE). The rate of each adverse event will be measured.

SECONDARY OUTCOMES:
Overall survival | From the beginning of the treatment to 2 years after the treatment.
  The time from the date of seeds implantation to the date of death from any cause or the date of last observation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: CSR
Time Frame: Data will be available within 6 month after the study completion.
Access Criteria: Data access requests will be reviewed by the research sponsor. Requestors will be required to sign a Data Access Agreement.